CLINICAL TRIAL: NCT01862835
Title: Impact of Estradiol Addback on Somatostatin Rebound in Older Men
Brief Title: Impact of Estradiol Addback
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13-000047
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Normal Healthy Volunteers
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Testosterone; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Degarelix/Te/placebo/ placebo (Experimental): Degarelix 80 mg (given as two s.c. injections of 60 mg) once [called day 1]; Te enanthate 100 mg i.m. given on day 1, 8 and 15; Oral placebo once daily x 22 days; and no patch beginning on day 1 and changed every 3 days through day 22.
  Interventions: Drug: Degarelix; Drug: Testosterone
- degarelix/Te/anastrozole/ placebo (Experimental): degarelix 80 mg (given as two s.c. injections of 60 mg) once [called day 1]; Te enanthate 100 mg i.m. given on day 1, 8 and 15; Oral anastrozole 2.0 mg once daily x 22 days; and no patch beginning on day 1 and changed every 3 days through day 22.
  Interventions: Drug: Degarelix; Drug: Testosterone; Drug: Anastrozole
- degarelix/Te/ anastrozole/E2 patch (Experimental): degarelix 80 mg (given as two s.c. injections of 60 mg) once [called day 1]; Te enanthate 100 mg i.m. given on day 1, 8 and 15; Oral anastrozole 2.0 mg once daily x 22 days; and an E2 patch calibrated to deliver 0.05 mg/day E2 beginning on day 1 and changed every 3 days through day 22.
  Interventions: Drug: Degarelix; Drug: Testosterone; Drug: Anastrozole; Drug: Estrogen patch
- degarelix/ placebo/placebo/no patch (Experimental): degarelix 80 mg (given as two s.c. injections of 60 mg) once [called day 1]; placebo i.m. given on day 1, 8 and 15; Oral placebo once daily x 22 days; and no patch beginning on day 1 and changed every 3 days through day 22.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix
Drug: Testosterone
  Arms: Degarelix/Te/placebo/ placebo; degarelix/Te/ anastrozole/E2 patch; degarelix/Te/anastrozole/ placebo
Drug: Anastrozole
  Arms: degarelix/Te/ anastrozole/E2 patch; degarelix/Te/anastrozole/ placebo
Drug: Estrogen patch
  Arms: degarelix/Te/ anastrozole/E2 patch

SUMMARY:
Repletion of testosterone (T) in older men drives Growth Hormone secretion after its aromatization to estradiol (E2) by potentiating endogenous GH drive.

DETAILED DESCRIPTION:
Systemic concentrations of Te, E2, GH, Insulin-like Growth Factor-I and IGFBP-3 decline in healthy aging men. Relative sex-steroid deprivation accentuates GH and IGF-I depletion, since Te stimulates GH and IGF-I production in older men, hypogonadal males of all ages, and patients undergoing (genotypic female-to-male) gender reassignment. Tamoxifen blocks this effect of Te, suggesting involvement of E2 in GH's stimulation in men. E2 per se stimulates GH secretion in women. Because Te is converted to E2 by aromatization in the body, we postulate that E2 is the active moiety in men also. Moreover, we hypothesize that the decline of E2 in older men contributes to the fall in GH output. This has never been tested. From a clinical vantage, understanding the mechanistic basis of Te's drive of the somatotropic axis is especially relevant in boys with pubertal failure, adults with primary hypogonadism and men with aging-related hypoandrogenemia. In relation to aging in the male, testosterone and E2 bioavailabilities fall by 35-50% in the eighth compared with third decade of life. From a medical perspective, aging is accompanied by progressive osteopenia, sarcopenia and intra-abdominal obesity. These adverse outcomes are remediable by short-term replacement with Te and/or recombinant GH, thus linking GH/Te/E2 availability with key body-compositional features.

ELIGIBILITY:
Inclusion:

* 60 healthy men (ages 60 to 80 y);
* BMI 18-30 kg/m2
* Community dwelling; and voluntarily consenting

Exclusion:

* Recent use of psychotropic or neuroactive drugs (within five biological half-live);
* Obesity (outside weight range above);
* Laboratory test results not deemed physician acceptable, cholesterol >250, triglycerides > 300, BUN >30 or creatinine > 1.5 mg/dL, liver functions tests twice upper limit of normal, electrolyte abnormality, anemia; hemoglobin <12.0 gm/dL
* Drug or alcohol abuse, psychosis, depression, mania or severe anxiety;
* Acute or chronic organ-system disease;
* Endocrinopathy, other than primary thyroidal failure receiving replacement; untreated osteoporosis
* Nightshift work or recent transmeridian travel (exceeding 3 time zones within 7 days of admission);
* Acute weight change (loss or gain of > 2 kg in 6 weeks);
* Allergy to peanut oil (used in some injectable Te preparations)
* Unwillingness to provide written informed consent.
* PSA > 4.0 ng/mL
* History or suspicion of prostatic disease (elevated PSA, indeterminate nodule or mass, obstructive uropathy.
* History of carcinoma (excluding localized basal cell carcinoma removed or surgically treated with no recurrence.
* History of thrombotic arterial disease (stroke, TIA, MI, angina) or deep vein thrombophlebitis.
* History of CHF, cardiac arrhythmias, congential QT prolongation, and medications used to treat cardiac arrhythmias
* Gynecomastia > 2 cm, untreated
* Untreated gallbladder disease
* History of smoking greater than one ppd.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
BioStatistical Analysis | Subjects will undergo 15-h overnight (2200 - 1300 h) fasting, 10-min blood sampling
  The primary analytical outcome is the summed mass of GH secreted in pulses over the 15 h of overnight blood sampling. The outcome measure is relevant, since sex-steroid hormones and regulatory peptides uniquely control GH secretory-burst mass.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Veldhuis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials